CLINICAL TRIAL: NCT01843075
Title: Evaluating the Effects of the Novel GLP-1 Analogue, Liraglutide, in Patients With Mild Alzheimer's Disease (ELAD Study)
Brief Title: Evaluating Liraglutide in Alzheimer's Disease
Acronym: ELAD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Imperial College London (Other)
Collaborators: King's College Hospital NHS Trust (Other); University of Oxford (Other); University of Southampton (Other); Avon and Wiltshire Mental Health Partnership NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: U1111-1131-9252
Record Dates: First submitted 2013-04-24; First posted 2013-04-30 (Estimated); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liraglutide (Experimental): Daily administration of 1.8 mg liraglutide by subcutaneous injection
  Interventions: Drug: Liraglutide
- Placebo (Placebo Comparator): Daily administration of matched placebo by subcutaneous injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Liraglutide — Daily subcutaneous injection
  Other Names: Victoza
  Arms: Liraglutide
Drug: Placebo — Daily subcutaneous injection
  Arms: Placebo

SUMMARY:
This is a 12-month, multicentre randomised double-blind placebo-controlled Phase IIb study in patients with mild Alzheimer's dementia (AD). Patients will be randomised on a 1:1 ratio to receive liraglutide or matching placebo.

DETAILED DESCRIPTION:
The investigators aim to recruit patients with mild Alzheimer's dementia as defined by the National Institute of Neurological and Communicative Disorders and Stroke - Alzheimer's Disease and Related Disorder Association (NINCDS-ADRDA) Criteria for Probable Alzheimer's Dementia or meeting Dubois criteria for early AD, with Mini Mental State Evaluation score of at least 20 out of a maximum of 30 and a CDR Global score of 0.5 or 1.

.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving and capacity to give informed consent
2. An individual who can act as a reliable study partner with regular contact (combination of face to face visits / telephone contact acceptable) who has sufficient subject interaction to provide meaningful input into rating scales and, if necessary, supervise or perform the injections, as judged by the investigator
3. Diagnosis of Probable Alzheimer's disease according to Dubois criteria (Dubois, Feldman et al. 2007) or National Institute of Neurological and Communicative Disorders and Stroke-Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria
4. Age from 50 years
5. Mini-Mental State Examination (MMSE) score of ≥20 and CDR-Global score of 0.5 or 1
6. Rosen Modified Hachinski Ischemic score ≤4
7. On stable medication for 2 months before the screening visit; on or off cholinesterase inhibitors
8. Fluency in English and evidence of adequate premorbid intellectual functioning
9. Likely to be able to participate in all scheduled evaluations and complete all required tests

Exclusion Criteria:

1. Patients on treatment for diabetes mellitus
2. Any contraindications to the use of liraglutide as per the Summary of Product Characteristics (hepatic impairment, renal impairment with CKD stage 4 and above (eGFR <30 ml/min/1.73m2), inflammatory bowel disease). Patients with eGFR less than 45 ml/min/1.73m2 will have the renal function monitored very closely
3. Significant neurological disease other than AD that may affect cognition
4. MRI/CT showing unambiguous aetiological evidence of cerebrovascular disease with regard to their dementia or vascular dementia fulfilling NINCDS-AIREN criteria
5. Current presence of a clinically significant major psychiatric disorder (e.g., Major Depressive Disorder) according to the criteria of the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV)
6. Current clinically significant systemic illness that is likely to result in deterioration of the patient's condition or affect the patient's safety during the study
7. History of epilepsy, where seizures or treatment could have contributed to cognitive impairment
8. Treatment with immunosuppressive medications (e.g. systemic corticosteroids) within the last 90 days (topical and nasal corticosteroids and inhaled corticosteroids for asthma are permitted) or chemotherapeutic agents for malignancy within the last 3 years
9. Myocardial infarction within the last 1 year
10. History of cancer within the last 5 years, except localised skin cancer
11. Other clinically significant abnormality on physical, neurological or laboratory examination that could compromise the study or be detrimental to the patient
12. History of alcohol or drug dependence or abuse within the last 2 years
13. Current use of anticonvulsant, anti-Parkinson's, anticoagulant (excluding the use of aspirin 325 mg/day or less) or narcotic medications. Subjects on anticoagulants will be allowed, but will not have an arterial line inserted
14. Use of experimental medications for AD or any other investigational medication or device within 60 days. Patients who have been involved in a monoclonal antibody study are excluded unless it is known that they were receiving placebo in that trial
15. Women of childbearing potential. Women who could become pregnant will be required to use adequate contraception throughout the trial
16. Patients with a personal or family history of medullary thyroid carcinoma (MTC) and patients with multiple endocrine neoplasia type 2 (MEN2)
17. Any contraindications to MRI scanning

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
The change in cerebral glucose metabolic rate | 12 months
  The change in cerebral glucose metabolic rate from baseline to follow up (12 months) in the treatment group compared with the placebo group.

SECONDARY OUTCOMES:
The change in z-scores for the ADAS Exec, MRI changes, microglial activation, and CSF markers | 12 months
  The change in z-scores for the ADAS Exec, MRI changes, microglial activation, and CSF markers
The incidence and severity of treatment emergent adverse events | 12 months
  The incidence and severity of treatment emergent adverse events or clinically important changes in safety assessments over 12 months.
The change in microglial activation | 12 months
  To establish whether there is a reduction in microglial activation in subjects with mild AD following daily subcutaneous injection of liraglutide for 1 year using TSPO PET scanning compared with subjects receiving placebo injections in a subgroup of patients
The change in tau deposition | 12 months
  The change in the hippocampal, entorhinal and other cortical changes in tau deposition in treatment group compared to the placebo group in a subgroup of subjects.
The change in cortical amyloid | 12 months
  Changes in levels of cortical amyloid load in treatment group compared to the placebo group in a subgroup of subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Edison, PhD FRCPI, Principal Investigator — Imperial College London
Locations (1):
- Imperial College, Hammersmith Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Edison P, Femminella GD, Ritchie C, Nowell J, Holmes C, Walker Z, Ridha B, Raza S, Livingston NR, Frangou E, Love S, Williams G, Lawrence R, Mcfarlane B, Archer H, Coulthard E, Underwood BR, Koranteng P, Karim S, Bannister C, Perneczky R, Prasanna A, Junaid K, McGuinness B, Nilforooshan R, Macharouthu A, Donaldson A, Thacker S, Russell G, Malik N, Mate V, Knight L, Kshemendran S, Holscher C, Mansouri A, Chester-Jones M, Holmes J, Tan T, Williams S, Ashraf A, Brooks DJ, Harrison J, Hinz R, Tadros G, Passmore AP, Ballard C. Liraglutide in mild to moderate Alzheimer's disease: a phase 2b clinical trial. Nat Med. 2026 Jan;32(1):353-361. doi: 10.1038/s41591-025-04106-7. Epub 2025 Dec 1. PMID 41326666
- [Derived] Femminella GD, Frangou E, Love SB, Busza G, Holmes C, Ritchie C, Lawrence R, McFarlane B, Tadros G, Ridha BH, Bannister C, Walker Z, Archer H, Coulthard E, Underwood BR, Prasanna A, Koranteng P, Karim S, Junaid K, McGuinness B, Nilforooshan R, Macharouthu A, Donaldson A, Thacker S, Russell G, Malik N, Mate V, Knight L, Kshemendran S, Harrison J, Holscher C, Brooks DJ, Passmore AP, Ballard C, Edison P. Evaluating the effects of the novel GLP-1 analogue liraglutide in Alzheimer's disease: study protocol for a randomised controlled trial (ELAD study). Trials. 2019 Apr 3;20(1):191. doi: 10.1186/s13063-019-3259-x. Erratum In: Trials. 2020 Jul 19;21(1):660. doi: 10.1186/s13063-020-04608-4. PMID 30944040
- [Derived] Muscogiuri G, DeFronzo RA, Gastaldelli A, Holst JJ. Glucagon-like Peptide-1 and the Central/Peripheral Nervous System: Crosstalk in Diabetes. Trends Endocrinol Metab. 2017 Feb;28(2):88-103. doi: 10.1016/j.tem.2016.10.001. Epub 2016 Oct 27. PMID 27871675